CLINICAL TRIAL: NCT03581058
Title: Investigating the Neural Correlates of Driving After Medical Cannabis Exposure
Brief Title: Neural Correlates of Driving and Cannabis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17-206
Record Dates: First submitted 2018-06-06; First posted 2018-07-10 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Cannabis Use; Driving Impaired
Keywords: MRI; Cannabis; Driving
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cannabis - Jean Guy (Experimental): A participant will be administered 1g of Jean Guy strain of cannabis.
  Interventions: Drug: Cannabis
- Cannabis - Churchill (Experimental): A participant will be administered 1g of Churchill strain of cannabis.
  Interventions: Drug: Cannabis
- Sober (No Intervention): All participants will complete same tasks sober.

INTERVENTIONS:
Drug: Cannabis — Participants will be assigned to consume one of the cannabis strains and will complete testing immediately after consumption.
  Other Names: Marijuana
  Arms: Cannabis - Churchill; Cannabis - Jean Guy

SUMMARY:
Driving is a set of complex tasks and requires use of multiple cognitive domains, including attention, planning, and memory. In laboratory studies, the main psychoactive component in cannabis, delta-9-tetrahydrocannabinol (THC), was shown to impair short-term memory, attention, reaction time, tracking, and coordination, resulting, for instance, in significantly more deviations from the lane and increased break latency. Surveys and epidemiological studies suggest that cannabis consumption is associated with increased risks of collision.

The current study aims to evaluate individual driving behavior and performance on various neurocognitive tests and their correlated neural networks while under the influence of cannabis and while sober. The investigators will use the STISIM driving simulator, which is fully MRI compatible, to study brain activation, while participants are performing various driving maneuvers.

The goals of the study are:

1. identify driving performance and patterns in brain activation associated with cannabis exposure and compare them to brain patterns of the same participants while sober;
2. compare participant's performance on cognitive tasks while under the influence of cannabis and sober;
3. look for correlations between concentration of cannabinoids in the participants' blood and their driving performance and performance on cognitive tasks;
4. correlate demographic variables and personal history (e.g. tolerance to drug) with performance and brain activation while driving under the influence of cannabis.

ELIGIBILITY:
Inclusion Criteria:

* valid driver's license
* have normal or corrected-to-normal vision
* have had prior experience consuming cannabis
* are currently not and have not been regular users in the past 5 years (regular use is defined as at least 1 time per week for at least 1 month)
* prescribed medical cannabis

Exclusion Criteria:

* not fluent in English
* do not meet MRI screening criteria
* use 50 mg/day of morphine equivalents
* history of neurological, neurodegenerative or psychiatric diseases
* any serious sensory or motor impairments
* pregnant women or women trying to get pregnant, or breastfeeding
* serious lung, liver, kidney, and heart problems, including angina, coronary artery disease, and arrhythmia, and Peripheral Vascular Disease
* personal or family history of mental disorders or alcohol or drug abuse or dependence

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in neural activation on fMRI during driving simulation | 30-60 min after cannabis intake vs sober
  Neural activation, based on BOLD signal, while completing driving tasks under the influence of cannabis and sober.

SECONDARY OUTCOMES:
Performance on driving simulator | 30-60 min after cannabis intake vs sober
  Number of errors while completing driving tasks (e.g. turning, driving straight, speed maintenance, missed stop signs, etc.) under the influence of cannabis and sober.
Performance on cognitive tasks | 60-90 min after cannabis intake vs sober
  Cognitive test battery to assess various driving-related cognitive functions: attention, working memory, visual-spatial processing, processing speed, etc.
Blood plasma concentration levels of cannabinoids | 10 min and 60 min after cannabis intake
  Concentration levels of THC and CBD throughout the session duration

CONTACTS AND LOCATIONS:
Overall Officials: Tom Schweizer, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No